CLINICAL TRIAL: NCT01835262
Title: Low Dose Ketamine Versus Morphine for Moderate to Severe Pain in the Emergency Department: A Prospective, Randomized, Double-Blind Study
Brief Title: Low Dose Ketamine Versus Morphine for Moderate to Severe Pain in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/09/VA01; 12-09-VA01 (Other: Maimonides Medical Center IRB)
Record Dates: First submitted 2013-04-12; First posted 2013-04-18 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: pain; Ketamine; Emergency Medicine; morphine
MeSH Terms: conditions — Pain | interventions — Morphine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): Morphine Group -- Receiving morphine at 0.1 mg /kg given as IVP
  Interventions: Drug: Morphine
- Ketamine Group (Experimental): Ketamine Group - - Receiving ketamine at 0.3 mg/given as IVP
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Morphine — Morphine: 0.1 mg /kg given as IVP
  Arms: Morphine
Drug: Ketamine — Ketamine:0.3 mg/given as IVP
  Arms: Ketamine Group

SUMMARY:
The primary objectives of the study are to evaluate the efficacy of subdissociative dose intravenous ketamine compared with intravenous morphine in relieving acute pain in the ED. Secondary objectives will include the rate of adverse effects and need for rescue analgesia. The hypothesis is that intravenous administration of subdissociative dose ketamine at 0.3 mg/kg is superior to intravenous morphine at 0.1mg/kg in treating moderate and severe acute pain in patients presenting to the ED.

DETAILED DESCRIPTION:
Rationale: Opioids are traditionally accepted as a cornerstone of acute pain management in the Emergency Department (ED). Morphine is one of the most commonly used parenteral opioid analgesics whose initial dose of 0.1 mg/kg has been extensively researched and recommended for control of severe acute pain in the ED. However, intravenous administration of opioids is associated with thefollowing side effects: hypotension, respiratory depression, dizziness, pruritis and nausea. In addition, in patients with pre-existing renal and/or hepatic insufficiency, these effects may be pronounced and require interventions. Thus, the administration of an equipotent analgesic that does not cause hypotension and respiratory depression would enhance patient safety in the ED.

Ketamine is a noncompetitive N-methyl D-aspartate (NMDA) receptor antagonist that blocks the release of excitatory neurotransmitter glutamate and provides anesthesia, amnesia and analgesia by virtue of decreasing central sensitization and "wind-up" phenomenon. Due to its high lipid solubility, ketamine rapidly crosses the blood-brain barrier, provides rapid onset of action (peak concentration at is reached 1 minute after IVP) and rapid recovery to baseline (duration of action 5-15 minutes after IVP) (1). When given at subdissociative doses of 0.1-0.5 mg/kg, either as an adjunct to opioid analgesic or as a solo agent, ketamine provides good analgesia while preserving airway patency, ventilation, and cardiovascular stability (2). In addition, a small dose of ketamine may increase the analgesic potency of opioids thus decreasing their dosing requirements (3). Based on the aforementioned facts, ketamine offers an attractive option for providing safe and convenient pain control for patients in the ED.

A double-blind trial of 40 adult patients with acute musculoskeletal trauma compared low-dose ketamine administered by subcutaneous infusion (0.1 mg/kg/h) with intermittent intravenous morphine (0.1 mg/kg IV every 4 hours ) and demonstrated better pain relief, less sedation and less nausea and vomiting with ketamine infusion than with intermittent morphine. In addition, none of the patients in the ketamine group required supplementary analgesia (4). A prospective, randomized trial compared two analgesic regimens, morphine with ketamine (K group) or morphine with placebo (P group) for severe acute pain in 73 trauma patients with a visual analog scale (VAS) score of at least 60/100. Morphine was administered at 0.1mg/kg; patients in the K group received 0.2 mg/kg of intravenous ketamine over 10 minutes while patients in the P group received isotonic sodium chloride solution. The results showed comparable change in VAS score at 30 minutes (34 mm (K) vs. 39 mm (P)) but reduced morphine consumption in the ketamine group (0.14 mg/kg (K) vs 0.2 mg/kg (P)) (5).

A chart review analysis of 35 ED patients receiving low dose ketamine at doses 0.1mg-0.6mg/kg in addition to intravenous morphine demonstrated a decrease in pain intensity for 54% of the patients by a documented 3 point pain decrease on a 10-point scale. The ketamine doses ranged from 5 mg to 35 mg with median dose of 10 mg and mean dose of 15.7mg. In addition, only one patient had a brief dysphoric reaction that did not require intervention (6).

Hypothesis: Intravenous administration of subdissociative dose ketamine at 0.3 mg/kg is superior to intravenous morphine at 0.1 mg/kg in treating moderate and severe acute pain in patients presenting to the ED.

Methods: Prospective, randomized, double-blind trial evaluating and comparing analgesic effect of intravenous Ketamine administered in sub-dissociative doses: 0.3 mg/kg given over 10 minutes with intravenous Morphine given at 0.1mg/kg as a single IVP.

Description: Once patient is triaged, an initial pain score will be assessed and patient's stated weight will be recorded in the chart. Patients will then have an initial evaluation by an attending ED physician and once found to be eligible for the study (deemed by treating physician to warrant administration of intravenous analgesia) patient will be randomized to receive either morphine at 0.1 mg /kg given as IVP or ketamine at 0.3 mg/given as IVP. Patients' vital signs will be recorded at triage, at the beginning of the study and at 15, 30, 60, 90, 120 minutes post-administration. Patients will be placed on a monitor and continuous pulse oximetry (oxygen saturation), blood pressure, heart rate and respiratory rate will be recorded. We will compare efficacy as a difference between 2 groups in pain relief from the baseline (at triage) to 30 minutes post-analgesic administration. The primary outcome is the difference between 2 groups in pain relief at 30 minutes. The secondary outcome is side effects. We will compare the safety profile of each analgesic with respect to incidence of hypotension, respiratory depression, nausea and vomiting, pruritis, need for an opioid reversal agent (naloxone), tachycardia, laryngospasm, hypersalivation, dizziness, agitation and need for benzodiazepines (midazolam) administration for symptomatic evidence of emergence reaction. All the data will be entered and analyzed via SPSS. Data analyses will include frequency distributions, and ANOVA to assess a difference in pain scores between the groups at various time points. All patients will be analyzed with an intent to treat analysis. However, a subgroup analysis will be done for any emergence reaction or event which occurs often.

ELIGIBILITY:
Inclusion Criteria:

1. ED patients18-55 years old presenting with moderate to severe (Numeric Pain Rating Score >5) acute (less than 7 days)
2. abdominal, flank, back or musculoskeletal pain warranting (in the treating physician's judgment) administration of intravenous opioid pain medication.
3. Patients must be awake, alert and oriented to time, place and person,
4. patient must be able to demonstrate understanding of the informed consent.
5. Patient must be able to verbalize how much pain they are having on the 10 point Numeric Rating Pain Scale,
6. Patient mus be able to verbalize the nature of the side effects he may be experiencing from the intravenous analgesia.

Exclusion Criteria:

1. Pregnancy or breast feeding
2. SBP<90
3. Weight greater than 115kg or less than 45kg,
4. altered mental status,
5. allergy to ketamine or morphine,
6. history of acute head or ocular trauma
7. presence of intracranial mass or vascular lesion, presence of psychiatric history
8. diagnosis or treatment (as assessed by electronic chart review).
9. history of seizure or intracranial hypertension
10. history of chronic pain, pain syndrome or fibromyalgia
11. presence of cardiovascular disease except controlled hypertension
12. history of acute head or ocular trauma, drug or alcohol abuse in the preceding 6 months
13. drugs or alcohol abuse in the preceding 6 months
14. SBP>180
15. HR<50
16. HR>150
17. RR<10
18. RR>30
19. administration of opiate pain medication in the past 4 hours prior to assessment (i.e. home, EMS, triage, office, etc.)
20. presence of renal or hepatic insufficiency (as assessed by electronic chart review),

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winterfield RW, Fadly AM, Hoerr FJ. Vaccination and revaccination with a Holland (H) strain of infectious bronchitis virus. Avian Dis. 1976 Apr-Jun;20(2):369-74. PMID 180959
- [Background] Javery KB, Ussery TW, Steger HG, Colclough GW. Comparison of morphine and morphine with ketamine for postoperative analgesia. Can J Anaesth. 1996 Mar;43(3):212-5. doi: 10.1007/BF03011736. PMID 8829857
- [Background] Gurnani A, Sharma PK, Rautela RS, Bhattacharya A. Analgesia for acute musculoskeletal trauma: low-dose subcutaneous infusion of ketamine. Anaesth Intensive Care. 1996 Feb;24(1):32-6. doi: 10.1177/0310057X9602400106. PMID 8669651
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Lester L, Braude DA, Niles C, Crandall CS. Low-dose ketamine for analgesia in the ED: a retrospective case series. Am J Emerg Med. 2010 Sep;28(7):820-7. doi: 10.1016/j.ajem.2009.07.023. Epub 2010 Apr 2. PMID 20837262

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine | Ketamine Group
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Ketamine Group | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.5) | 34.8 (9.5) | 35.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90
Numeric Rating Scale of Pain score [Mean (Standard Deviation); unit: score] — Numeric Rating Scale of Pain Score (0=no pain and 10=severe pain)
  score | 8.49 (1.5) | 8.64 (1.5) | 8.57 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale of Pain
Description: We will compare efficacy as a difference between 2 groups in pain score at 30 minutes post-analgesic administration. The primary outcome is the difference between 2 groups in pain score at 30 minutes.
  Pain will be measured via Numeric rating scale from 0 to 10 with 0 being no pain, 5 being moderate pain, and 10 being severe pain
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Morphine | Ketamine Group
Number analyzed (Participants) | 45 | 45
Units on a scale | 3.93 (3.1) | 4.07 (3.2)

ADVERSE EVENTS:
Time Frame: Within 2 hours of administration of either morphine or ketamine
Arm/Group | Morphine | Ketamine Group
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 15/45 | 14/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=45) | Ketamine Group (N=45)
Dizziness (General disorders) | 6 (6) | 8 (8) — Dizziness
Nausea (Gastrointestinal disorders) | 9 (9) | 6 (6) — Nausea

LIMITATIONS AND CAVEATS:
This was a single center study in which patients were enrolled as a convenience. There was the potential for unblinding as some participants exhibited ketamine specific reactions such as nystagmus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes